CLINICAL TRIAL: NCT00089570
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Phase III Study of Intravenous Terlipressin in Patients With Hepatorenal Syndrome Type 1
Brief Title: Study of Terlipressin Versus Placebo to Treat Hepatorenal Syndrome Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OT-0401
Record Dates: First submitted 2004-08-06; First posted 2004-08-09 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Hepatorenal Syndrome
Keywords: hepatorenal syndrome; terlipressin
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Terlipressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Terlipressin (Experimental): Terlipressin
  Interventions: Drug: terlipressin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: terlipressin
  Arms: Terlipressin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether terlipressin is safe and effective in the treatment of patients with hepatorenal syndrome (HRS) type 1 when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, or acute liver disease
* Rapidly progressive reduction in renal function, e.g. doubling of serum creatinine to >2.5 mg/dL in less than two weeks.
* No sustained improvement in renal function after diuretic withdrawal and plasma volume expansion
* Proteinuria <500 mg per day
* No evidence of granular casts in urinalysis or ultrasonographic evidence of obstructive uropathy or parenchymal renal disease

Exclusion Criteria:

* Ongoing shock
* Uncontrolled bacterial infection
* Current significant fluid losses
* Current or recent treatment with nephrotoxic drugs (e.g. NSAIDs or aminoglycosides within 4 weeks)
* Acute liver disease due to factors known to be also directly nephrotoxic (e.g. acetaminophen overdose)
* Confirmed pregnancy
* Severe cardiovascular disease
* Evidence of intrinsic or parenchymal renal disease (e.g. acute tubular necrosis)
* Participation in other clinical studies within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Treatment Success | Day 14

SECONDARY OUTCOMES:
Renal function and survival | Renal funtion to Day 14 and Survival to Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Arun J. Sanyal, M.D., Study Chair — Medical College of Virginia, Virginia Commonwealth University Medical Center; Thomas D. Boyer, M.D., Study Director — University of Arizona Health Sciences Center; Peter Teuber, Ph.D., Study Director — Orphan Therapeutics
Locations (37):
- United States (37):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Arizona College of Medicine, Tucson, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCSD Medical Center Hillcrest, San Diego, California
  - VA Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Hospital & Health Sciences Center, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - VA CT Health Care System, West Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Fairview-University Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - 983285 Nebraska Medical Center, Omaha, Nebraska
  - University of Medicine & Dentistry of New Jersey - NJMS, Newark, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Mount Sinai Medical Center/Mount Sinai Hospital, New York, New York
  - Center for Liver Disease & Transplantation Clinic, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center of Dallas, Dallas, Texas
  - St. Luke's Episcopal Hospital, St. Luke's Texas Liver Institute, Houston, Texas
  - VCU Medical Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Background] Arroyo V, Guevara M, Gines P. Hepatorenal syndrome in cirrhosis: pathogenesis and treatment. Gastroenterology. 2002 May;122(6):1658-76. doi: 10.1053/gast.2002.33575. No abstract available. PMID 12016430
- [Background] Colle I, Durand F, Pessione F, Rassiat E, Bernuau J, Barriere E, Lebrec D, Valla DC, Moreau R. Clinical course, predictive factors and prognosis in patients with cirrhosis and type 1 hepatorenal syndrome treated with Terlipressin: a retrospective analysis. J Gastroenterol Hepatol. 2002 Aug;17(8):882-8. doi: 10.1046/j.1440-1746.2002.02816.x. PMID 12164964
- [Background] Duhamel C, Mauillon J, Berkelmans I, Bourienne A, Tranvouez JL. Hepatorenal syndrome in cirrhotic patients: terlipressine is a safe and efficient treatment; propranolol and digitalic treatments: precipitating and preventing factors? Am J Gastroenterol. 2000 Oct;95(10):2984-5. doi: 10.1111/j.1572-0241.2000.03214.x. No abstract available. PMID 11051385
- [Background] Hadengue A, Gadano A, Moreau R, Giostra E, Durand F, Valla D, Erlinger S, Lebrec D. Beneficial effects of the 2-day administration of terlipressin in patients with cirrhosis and hepatorenal syndrome. J Hepatol. 1998 Oct;29(4):565-70. doi: 10.1016/s0168-8278(98)80151-7. PMID 9824265
- [Background] Halimi C, Bonnard P, Bernard B, Mathurin P, Mofredj A, di Martino V, Demontis R, Henry-Biabaud E, Fievet P, Opolon P, Poynard T, Cadranel JF. Effect of terlipressin (Glypressin) on hepatorenal syndrome in cirrhotic patients: results of a multicentre pilot study. Eur J Gastroenterol Hepatol. 2002 Feb;14(2):153-8. doi: 10.1097/00042737-200202000-00009. PMID 11981339
- [Background] Moreau R, Durand F, Poynard T, Duhamel C, Cervoni JP, Ichai P, Abergel A, Halimi C, Pauwels M, Bronowicki JP, Giostra E, Fleurot C, Gurnot D, Nouel O, Renard P, Rivoal M, Blanc P, Coumaros D, Ducloux S, Levy S, Pariente A, Perarnau JM, Roche J, Scribe-Outtas M, Valla D, Bernard B, Samuel D, Butel J, Hadengue A, Platek A, Lebrec D, Cadranel JF. Terlipressin in patients with cirrhosis and type 1 hepatorenal syndrome: a retrospective multicenter study. Gastroenterology. 2002 Apr;122(4):923-30. doi: 10.1053/gast.2002.32364. PMID 11910344
- [Background] Mulkay JP, Louis H, Donckier V, Bourgeois N, Adler M, Deviere J, Le Moine O. Long-term terlipressin administration improves renal function in cirrhotic patients with type 1 hepatorenal syndrome: a pilot study. Acta Gastroenterol Belg. 2001 Jan-Mar;64(1):15-9. PMID 11322061
- [Background] Solanki P, Chawla A, Garg R, Gupta R, Jain M, Sarin SK. Beneficial effects of terlipressin in hepatorenal syndrome: a prospective, randomized placebo-controlled clinical trial. J Gastroenterol Hepatol. 2003 Feb;18(2):152-6. doi: 10.1046/j.1440-1746.2003.02934.x. PMID 12542598
- [Background] Suzuki H, Stanley AJ. Current management and novel therapeutic strategies for refractory ascites and hepatorenal syndrome. QJM. 2001 Jun;94(6):293-300. doi: 10.1093/qjmed/94.6.293. PMID 11391027
- [Background] Uriz J, Gines P, Cardenas A, Sort P, Jimenez W, Salmeron JM, Bataller R, Mas A, Navasa M, Arroyo V, Rodes J. Terlipressin plus albumin infusion: an effective and safe therapy of hepatorenal syndrome. J Hepatol. 2000 Jul;33(1):43-8. doi: 10.1016/s0168-8278(00)80158-0. PMID 10905585
- [Derived] Bajaj JS, Kwo P, Pappas SC, O'Leary JG, Jamil K, Cardoza S, Wong F. Bradycardia and Other Arrhythmias in Patients With Hepatorenal Syndrome-Acute Kidney Injury Following Terlipressin Treatment: A Pooled Analysis of Three North American Phase III Clinical Studies. Aliment Pharmacol Ther. 2025 Dec;62(11-12):1192-1201. doi: 10.1111/apt.70297. Epub 2025 Jul 24. PMID 40704461
- [Derived] Mujtaba MA, Gamilla-Crudo AK, Merwat SN, Hussain SA, Kueht M, Karim A, Khattak MW, Rooney PJ, Jamil K. Terlipressin in combination with albumin as a therapy for hepatorenal syndrome in patients aged 65 years or older. Ann Hepatol. 2023 Sep-Oct;28(5):101126. doi: 10.1016/j.aohep.2023.101126. Epub 2023 Jun 10. PMID 37302573
- [Derived] Velez JCQ, Wong F, Reddy KR, Sanyal AJ, Vargas HE, Curry MP, Gonzalez SA, Pappas SC, Jamil K. The Effect of Terlipressin on Renal Replacement Therapy in Patients with Hepatorenal Syndrome. Kidney360. 2023 Aug 1;4(8):1030-1038. doi: 10.34067/KID.0000000000000132. Epub 2023 May 5. PMID 37143199
- [Derived] Curry MP, Vargas HE, Befeler AS, Pyrsopoulos NT, Patwardhan VR, Jamil K. Early treatment with terlipressin in patients with hepatorenal syndrome yields improved clinical outcomes in North American studies. Hepatol Commun. 2023 Jan 3;7(1):e1307. doi: 10.1097/01.HC9.0000897228.91307.0c. eCollection 2023 Jan 1. PMID 36633470
- [Derived] Sanyal AJ, Boyer TD, Frederick RT, Wong F, Rossaro L, Araya V, Vargas HE, Reddy KR, Pappas SC, Teuber P, Escalante S, Jamil K. Reversal of hepatorenal syndrome type 1 with terlipressin plus albumin vs. placebo plus albumin in a pooled analysis of the OT-0401 and REVERSE randomised clinical studies. Aliment Pharmacol Ther. 2017 Jun;45(11):1390-1402. doi: 10.1111/apt.14052. Epub 2017 Mar 29. PMID 28370090
- [Derived] Sanyal AJ, Boyer T, Garcia-Tsao G, Regenstein F, Rossaro L, Appenrodt B, Blei A, Gulberg V, Sigal S, Teuber P; Terlipressin Study Group. A randomized, prospective, double-blind, placebo-controlled trial of terlipressin for type 1 hepatorenal syndrome. Gastroenterology. 2008 May;134(5):1360-8. doi: 10.1053/j.gastro.2008.02.014. Epub 2008 Feb 13. PMID 18471513